CLINICAL TRIAL: NCT06664944
Title: Technology Exposure and Child Health: Wellness Impact and Social Effects (TECHWISE): an Observational Product Registry Study
Brief Title: Technology Exposure and Child Health: Wellness Impact and Social Effects: an Observational Product Registry Study
Acronym: TECHWISE
Status: Recruiting | Type: Observational
Sponsor: Aura (Industry)
Responsible Party: Sponsor
Other Study IDs: 20243405
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-10

CONDITIONS: Mood; Depression Disorders; Anxiety Disorders; Sleep; Eating Disorders; Physical Activity; Loneliness; Stress
Keywords: digital health; digital mental health; technology impacts on mental health; digital natives; digital parenthood; child online safety; digital wellness; child online well-being
MeSH Terms: conditions — Anxiety Disorders; Feeding and Eating Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children 8-17 years old: Over 84% of children ages 8 and up have access to a mobile device (smartphone, tablet) and are active on social media. This study focuses on children ages 8-17 to better understand social media usage and how it relates to their mental well-being.

SUMMARY:
The goal of this study is to understand how children's mobile device usage (smartphones or tablets), including social media use and online games, are related to their mental wellness and mental health, as well as some aspects of their physical activity and sleep. This study is available to all children between the ages of 8 and 17 years and a parent/caregiver.

Researchers will compare participant mobile device usage with their survey responses on sleep, stress, mental health, and physical activity, as well as their parent/caregiver's survey responses.

Participants will:

* run the Aura app with parental controls on their dedicated mobile device
* complete monthly surveys
* answer daily questions on mood, stress, sleep and physical activity

The study is fully virtual. Duration is 3 months.

DETAILED DESCRIPTION:
Once enrolled, child participants will use their mobile devices as usual, and Aura will collect data on on-line and off-line activity, app usage, social interaction, sleep, location and activity levels.

The child participant will complete surveys on a monthly basis, including:

* A range of questionnaires about feelings and behaviors that are associated with mental health challenges
* Questionnaires that ask about well-being and positive feelings, including relationships with family and friends
* Questionnaires that ask about experiences with social media and device usage
* A questionnaire about feelings of loneliness
* A questionnaire that asks about activity sleep

In parallel, the parent participant will complete monthly surveys about the child, including:

* Medical history and changes
* A range of questionnaires about feelings and behaviors that are associated with mental health challenges
* Questionnaires that ask about well-being and positive feelings, including relationships with family and friends

ELIGIBILITY:
Inclusion Criteria:

1. Child participants are male, female, non-binary persons, ages 8-17, inclusive
2. Parent/Authorized Legal Guardian willing to provide informed consent; child willing to provide assent
3. Both Parent/Authorized Legal Guardian and child own a mobile device that already has the Aura app or is able to install and run the Aura app, and the appropriate parental control features.
4. Parent/Authorized Legal Guardian and child are willing for child to use a dedicated device for the duration of the study (ie., child cannot share device with a sibling or other family member).
5. Multiple children from the same family are eligible to participate, provided that each enrolled child uses a dedicated device AND is able to complete outcome assessments independently, AND that parent/authorized legal guardian is able to complete assessments for each enrolled child.
6. Both Parent/Authorized Legal Guardian and child willing to share data collected as part of the Aura app and related device applications
7. Consented Parent/Authorized Legal Guardian and child maintain active Aura accounts throughout their study participation
8. Consented Parent/Authorized Legal Guardian and child are able to follow written and verbal instructions (English) as assessed by the PI and/or study coordinator
9. Consented Parent/Authorized Legal Guardian and child are to comply with all testing and study requirements

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: US-based, English-speaking, parents and children who use mobile devices for social media and online games.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assess ongoing technology use to explore children's online behaviors and derived health behaviors. | December 2025
  Assess ongoing technology use via the Aura app, including social media and other online behaviors, as well as other smartphone derived health behaviors, such as sleep, location, and activity levels.

SECONDARY OUTCOMES:
Examine bivariate associations between technology use features and mental wellness and mental health outcomes | December 2025
  Given the wide range of variables that can be derived from the Aura app, and the number of assessments that will be collected, all analyses should be considered exploratory. As an initial exploration of this objective, we will conduct simple bivariate analyses between technology use variables and mental health outcomes. Example questions include:
  * Are the temporal patterns of device usage (eg., more evening or late-night use) associated with sleep or physical activity outcome measures?
  * Does digital stress mediate the relationship between device usage and mental health outcomes?
Develop preliminary predictive models that use technology use and smartphone-derived parameters to predict point-in-time mental health outcomes | December 2025
  Develop preliminary predictive models that use technology use and smartphone-derived parameters to predict point-in-time mental health outcomes, as well as change over time.
  A wide range of analytic techniques will be used to develop and evaluate predictive models to determine whether mental health related outcomes and their change over time can be reliably predicted from device usage data. Example prediction models that may be evaluated but are not limited to the following:
  Do patterns/changes in device-mediated social interactions predict presence/severity of loneliness? Are there specific patterns of keyboard data (specific search terms, text messaging sentiment, etc.) that predict changes in mood or anxiety outcomes? Related, do patterns of keyboard activity map onto daily ratings of mood/stress/anxiety? Can patterns of device usage predict changes in health care utilization over time?

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kollins, Doctorate in Psychology, Principal Investigator — Aura
Locations (1):
- Aura, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kollins SH, Flannery J, Goetz K, Akre-Bhide S. Technology Effects and Child Health: Wellness Impact and Social Effects (TECHWISE): Protocol for a Prospective, Observational, Real-World Study. JMIR Res Protoc. 2025 Jun 19;14:e69358. doi: 10.2196/69358. PMID 40424191